CLINICAL TRIAL: NCT06240650
Title: Randomized Controlled Study to Evaluate Tolerability of a Modified Health-Dx
Brief Title: Tolerability of a Modified Health-Dx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celero Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEL-005
Record Dates: First submitted 2023-12-28; First posted 2024-02-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- modified Health- Dx™ (mHDx) study capsule (Experimental)
  Interventions: Device: modified Health- Dx™ (mHDx) study capsule
- modified Health- Dx™ (mHDx) control capsule (Other)
  Interventions: Device: modified Health- Dx™ (mHDx) control capsule

INTERVENTIONS:
Device: modified Health- Dx™ (mHDx) study capsule — The Study mHDx capsule has a mechanism that allows the mHDx to remain resident in the stomach for no more than six (6) hours. After this residency period, the Study mHDx will disassemble and pass safely through the subject's gastrointestinal system.
  Arms: modified Health- Dx™ (mHDx) study capsule
Device: modified Health- Dx™ (mHDx) control capsule — The Control mHDX capsule does not have a functional residency mechanism so it will disassemble once safely through the esophagus (within 10 minutes) and will then pass safely through the subject's gastrointestinal system.
  Arms: modified Health- Dx™ (mHDx) control capsule

SUMMARY:
Single Blind, Randomized Control Study is designed to evaluate the tolerability of the Celero Systems' modified Health-Dx™ (mHDx) capsule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals ages 18 - 75 inclusive
* Subject is a suitable candidate for study participation in the opinion of the Investigator
* Subject has been informed of the nature of the study and has provided written informed consent as approved by the WVU IRB

Exclusion Criteria:

* Subjects with a history of any condition that may impact the GI tract
* Subjects who are unable to swallow a 000 sized capsule
* Subjects with an implanted medical device that has wireless data communication capability
* Subjects planning to undergo an MRI within 30 days after the study
* Subjects with a BMI > 40 (severe obesity)
* Subjects who are pregnant or are nursing
* Any subject deemed to be at risk of a gastrointestinal complication as evaluated by a gastroenterologist prior to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
The difference, if any, in tolerability between the Study and Control as reported via the study questionnaire. mHDx as reported by the subjects. | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No